CLINICAL TRIAL: NCT06017193
Title: Ultrasonic Imaging of Bone Graft Healing in Extraction Sockets for Precise and Personalized Implant Therapy (HUM00226516)
Brief Title: Ultrasound for Socket Healing Evaluation
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Oliver Kripfgans, Associate Professor, University of Michigan
Other Study IDs: HUM00226516; 1R01DE030872 (NIH)
Record Dates: First submitted 2023-08-01; First posted 2023-08-30 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Healing Wound; Alveolar; Wound; Alveolar Bone Loss; Image; Dent Disease
MeSH Terms: conditions — Wounds and Injuries; Alveolar Bone Loss; Dent Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue core biopsy from healed sockets.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The design is a single blinded, dual comparative study of ultrasound versus micro-CT/LASCA in one study group. Up to a total of 140 subjects registered will be recruited. Subjects who are treatment planned for extraction of a hopeless tooth and socket augmentation with bone graft and are planned for a dental implant surgery. The socket will be evaluated before the extraction and multi-time points during healing until an implant is placed with various evaluation tools, including ultrasound.

DETAILED DESCRIPTION:
The design is a single blinded, dual comparative study of ultrasound versus micro-CT/LASCA in one study group. Up to a total of 140 subjects registered will be recruited. Subjects who are treatment planned for extraction of a hopeless tooth and socket augmentation with bone graft and are planned for a dental implant surgery. Qualified subjects will be asked during their pre-assessment visit. Subjects will be scanned with ultrasound and LASCA among other assessments shown in the info-graph and schedule of events. At the day of tooth extraction and socket augmentation (graft placement), clinical exams/measurements are taken, along with other research activities described in the info-graph and schedule of events. Recovery (checkups) from surgery will be monitored at 2 weeks, 1 month and 2 months, and 3 months. The timepoints additional to normal clinical timepoints are needed to gather potentially diagnostic valuable information about graft maturation, which in the future may lead to an early graft failure decision or trigger other clinical steps such as infection management.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age and have at least a tooth that is considered hopeless, planned for an extraction and a bone grafting procedure for subsequent dental implant surgery.

Exclusion Criteria:

* Patients not willing or not able to have an extraction, bone graft and subsequent implant surgery due to health, finance, or any other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who are treatment planned for extraction of a hopeless tooth and socket augmentation with bone graft and are planned for a dental implant surgery.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | approximately 6 months
  To determine if bone graft maturation can be imaged by ultrasound. Bone healing by ultrasound will be given a scale and will be compared to the reference standard micro-computed tomography (micro-CT) of tissue core biopsy taken at implant surgery

SECONDARY OUTCOMES:
Secondary Objective | approximately 6 months
  To determine if bone graft maturation can be imaged by ultrasound, by comparing to clinical healing appearances. A score will be given to ultrasound image and clinical outcome and the correlation will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Kripfgans, PhD, Principal Investigator — University of Michigan, Radiology
Locations (1):
- Ohio State University, Columbus, Ohio, United States